CLINICAL TRIAL: NCT01392391
Title: Jamaica and Maryland Mobility in Stroke
Brief Title: Exercise For Sub-acute Stroke Patients in Jamaica
Acronym: JAMMS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Rich Macko, MD, Baltimore VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00048469; R01HD068712 (NIH)
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Stroke
Keywords: Stroke; Exercise; Protein synthesis; Protein breakdown; Muscle atrophy; Muscle phenotype; Inflammation; Insulin resistance; Fitness
MeSH Terms: conditions — Stroke; Motor Activity; Muscular Atrophy; Inflammation; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): Task-oriented exercise training (aerobic, strength, and balance exercises)
  Interventions: Procedure: Task Oriented Exercise Training
- Stroke Care (Active Comparator): Best Medical Care in Jamaica adapted from the American Stroke Association "Get with the Guidelines".
  Interventions: Procedure: Stroke Care "Get with the Guidelines"

INTERVENTIONS:
Procedure: Task Oriented Exercise Training — Treadmill training with safety harnesses begin at 6 to 15 minutes total duration at 40-50% maximal heart rate reserve 3 times per week, increasing to 60-70% maximal heart rate reserve for 30 minutes for 6 months.
  Group dynamic balance exercise immediately follow the treadmill training 3 times a week. Participants also receive Best Stroke Care according to "Get with the Guidelines"
  Arms: Exercise
Procedure: Stroke Care "Get with the Guidelines" — Post-stroke care is applied according to the recommendations of the American Stroke Association "Get with the Guidelines" adapted for Jamaica
  Arms: Stroke Care

SUMMARY:
Chronic hemiparetic stroke is associated changes in body composition, skeletal muscle and cardiometabolic health; specific changes include paretic limb muscular atrophy, increased intramuscular fat deposition, elevated prevalence of impaired glucose tolerance and type 2 diabetes. This randomized intervention study compares a 6 month task oriented exercise programs versus control with both groups receiving best medical stroke care according to American Stroke Association "Get with the Guidelines". The hypothesis is that is 6 months of task-oriented exercise initiated early across the sub-acute period of stroke can prevent or ameliorate the natural course of these body composition, skeletal muscle and cardiometabolic health changes.

DETAILED DESCRIPTION:
Stroke leads to profound cardiovascular deconditioning and secondary abnormalities in paretic skeletal muscle that worsen cardiovascular health. Conventional rehabilitation focuses on restoration of daily function, without an adequate exercise stimulus to address deconditioning or the muscle abnormalities that may propagate insulin resistance (IR) to worsen risk for type 2 diabetes mellitus (T2DM) and recurrent stroke. By the time individuals reach chronic stroke (>6 months), we report hemiparetic body composition abnormalities including paretic leg muscular atrophy, increased intramuscular area fat, and a major shift to fast myosin heavy chain (MHC). All of these factors promote IR, which has been linked to reduced muscle protein synthesis in aging that may be reversible with exercise. We also find elevated tumor necrosis factor alpha (TNFα) in paretic leg muscle, suggesting that inflammation may affect protein synthesis and breakdown, similar to sarcopenia in aging. Yet, no prior studies have considered stroke as a catabolic syndrome modifiable by early exercise to improve muscle and cardiometabolic health.

Aim #1. Paretic (P) and non-paretic (NP) leg mixed muscle protein synthesis and breakdown in the fed and fasted state, TNFα expression, thigh muscle volume and strength.

Hypothesis 1: Paretic leg has reduced muscle protein synthesis and increased breakdown compared to non-paretic leg; TEXT will increase mixed muscle protein synthesis and reduce breakdown to increase muscle volume and strength by the mechanism(s) of reducing inflammation in the paretic leg, compared to controls.

Aim # 2. Glucose tolerance, fitness, and muscle phenotype. Hypothesis 2: TEXT will improve fitness levels, insulin and glucose response to oral glucose challenge, and increase paretic leg slow twitch (slow MHC) muscle molecular phenotype.

This randomized study investigates the hypothesis that in African-Jamaican adults with recent hemiparetic stroke, 6 months of TEXT across the sub-acute and into the chronic phase of stroke will improve paretic leg muscle and cardiometabolic health, compared to controls receiving best medical care.

Phase 1 consists of recruitment and screening of individuals with mild to moderate hemiparetic stroke from UWI Accident and Emergency Room and Neurology Stroke Clinics. Phase 2: Subjects with hemiparetic gait ≤ 8 weeks post-stroke who are not wheelchair bound or bed are approached for informed consent, medical, neurologic, blood tests, and treadmill (TM) exercise tests to determine study eligibility. Phase 3 baseline testing includes measures of fitness, oral glucose tolerance test (OGTT), body composition, bilateral vastus lateralis muscle biopsies, stable isotope measures of protein synthesis and breakdown. Phase 4: Eligible subjects are randomized to 6 months 3x/week TEXT or control group with best medical care alone that includes American Stroke Association (ASA) physical activity guideline recommendations for walking 4x/week. Randomization is stratified based on glucose tolerance (normal vs. abnormal) and gait deficit severity. Subjects have limited 3 month testing of fitness levels (VO2 peak), body composition, fasting glucose and insulin levels to document the natural history (controls) and temporal profile of exercise-mediated adaptations (TEXT) as they transition from the sub-acute into chronic phase of stroke. Phase 5 is 6-month post-intervention testing.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke within 8 weeks
* BMI of 18-40 kg/m2
* Able to walk 3 minutes with handrails, assistive device, or standby aid

Exclusion Criteria:

* Actively exercising for >30 minutes per day for 5 days per week
* Increased alcohol consumption (> 2 oz. liquor, 8 oz. wine, 24 oz. beer per day)
* Active abuse of other illegal and illicit drugs
* Cardiac History of: a) unstable angina, b) recent (<3 months) myocardial infarction, congestive heart failure (NYHA category II-IV), c) hemodynamically significant valvular dysfunction
* Medical History: a) peripheral arterial disease with vascular claudication making exercise challenging, b) orthopedic or chronic pain condition(s) restricting exercise, c) pulmonary or renal failure, d) active cancer, e) untreated poorly controlled hypertension measured on at least 2 occasions (greater than 160/100), f) HIV-AIDS or other known inflammatory responses, g) sickle cell anemia, h) medications: heparin, warfarin, lovenox, or oral steroids, j) currently pregnant
* Endocrine History: a) type 1 diabetes or insulin dependent type 2 diabetes, b) poorly controlled type 2 diabetes (HbA1C > 10)
* Neurological History: a) dementia (Mini-Mental Status score < 23 or < 17 if education level at or below 8th grade) and clinical confirmation by clinical evaluation, b) severe receptive or global aphasia that confounds testing and/or training, operationally defined as unable to follow 2 point commands, c) hemiparetic gait from a prior stroke preceding the index stroke defining eligibility (more than one stroke), d) neurologic disorder restricting exercise such as Parkinsons or myopathy, e) untreated major depression (CESD > 16 or clinical confirmation), f) muscular disorder (s) restricting exercise
* Muscle biopsy exclusion criteria: a) anti-coagulation therapy with heparin, warfarin, or lovenox (anit-platelet therapy is permitted), b)bleeding disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-07; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Thigh and Abdominal muscle and fat | Baseline and 6 months
  CT scans to determine 1) mid-thigh cross sectional area for muscle area, intramuscular and subcutaneous fat area, and quality of lean tissue mass, 2) abdominal fat area.
Whole body protein and skeletal muscle synthesis and breakdown | Baseline and 6 months
  Serial blood sampling and pre-/post-muscle biopsies in the fasted and fed state
Muscle myosin heavy chain isoform (MHC) proportions | Baseline and 6 months
  Analysis of muscle biopsies for MHC fiber type proportions
Leg Strength | Baseline and 6 months
  1 repetitive maximum strength for leg extension, quadriceps and hamstring muscles
Fitness | Baseline and 6 months
  VO2 peak testing with open circuit spirometry
Glucose tolerance | Baseline and 6 months
  2 hour oral glucose tolerance test with serial blood sampling every 30 minutes for glucose and insulin

SECONDARY OUTCOMES:
Muscle TNF alpha | Baseline and 6 months
  Analysis of muscle biopsy samples for TNF levels
Mobility and balance | Baseline and 6 months
  Stroke deficit profile will be indexed by NIH Stroke Scale, modified Ashworth, timed walks, Short Physical Performance Battery, Berg Balance.

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Macko, MD, Principal Investigator — University of Maryland; Terrence Forrester, MD, Principal Investigator — University of West Indies
Locations (2):
- University of Maryland, Baltimore, Maryland, United States
- University of West Indies, Kingston, Mona 7, Jamaica

REFERENCES:
- [Background] Michael K, Goldberg AP, Treuth MS, Beans J, Normandt P, Macko RF. Progressive adaptive physical activity in stroke improves balance, gait, and fitness: preliminary results. Top Stroke Rehabil. 2009 Mar-Apr;16(2):133-9. doi: 10.1310/tsr1602-133. PMID 19581199
- [Background] Lam JM, Globas C, Cerny J, Hertler B, Uludag K, Forrester LW, Macko RF, Hanley DF, Becker C, Luft AR. Predictors of response to treadmill exercise in stroke survivors. Neurorehabil Neural Repair. 2010 Jul-Aug;24(6):567-74. doi: 10.1177/1545968310364059. Epub 2010 May 7. PMID 20453154
- [Background] Luft AR, Macko RF, Forrester LW, Villagra F, Ivey F, Sorkin JD, Whitall J, McCombe-Waller S, Katzel L, Goldberg AP, Hanley DF. Treadmill exercise activates subcortical neural networks and improves walking after stroke: a randomized controlled trial. Stroke. 2008 Dec;39(12):3341-50. doi: 10.1161/STROKEAHA.108.527531. Epub 2008 Aug 28. PMID 18757284
- See also: American Stroke Association — http://www.strokeassociation.org/STROKEORG/
- See also: University of West Indies Tropical Medicine Research Unit — http://www.uwi.edu/tmri/default.aspx